CLINICAL TRIAL: NCT03847740
Title: Safety and Feasibility of a New Neuromuscular Monitoring Device
Acronym: MONITOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MONITOF
Record Dates: First submitted 2019-01-21; First posted 2019-02-20 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: General Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right Isometric Thumb Force (ITF) handle (Experimental)
  Interventions: Device: Isometric Trumb Force handle
- Left Isometric Thumb Force (ITF) handle (Experimental)
  Interventions: Device: Isometric Trumb Force handle

INTERVENTIONS:
Device: Isometric Trumb Force handle — Compare the pattern of neuromuscular blocking drug between two devices applied on the same patient during general anesthesia.

SUMMARY:
The aim of the study is to compare, during general anesthesia using neuromuscular blocking agent, the feasibility of a new mechanographic device (ITF handle and Visual ITF software) with a standard acceleromyographic device (TOF Watch SX) and also to assess its safety during the first 24 hours after surgery.

The two devices will be studied simultaneously in each patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients,
* ASA class 1 to 3,
* Scheduled for elective surgery requiring general anesthesia and muscle paralysis

Exclusion Criteria:

* Age inferior to 18 years,
* ASA class 4,
* Emergency surgery,
* Prone position on the operating table

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Delay of block installation between the injection and the disappearance of all the muscular contractions to stimulation by train of four | Usefulness of non depolarizing muscle relaxant-induced muscle paralysis is limited at the surgery period and should be avoided once the surgery is completed. Therefore, all measurements are done during this time.
  We compare the response to curare with one side a conventional TOF Watch SX monitor and other side Handle Isometric Thumb Force.

SECONDARY OUTCOMES:
Clinical examination | the first 24 postoperative hours
  Appearance of the wrist skin (for example: redness, irritations or marks)
Clinical examination | the first 24 postoperative hours
  Wrist pain
Characteristics of maintenance curarization | Usefulness of non depolarizing muscle relaxant-induced muscle paralysis is limited at the surgery period and should be avoided once the surgery is completed. Therefore, all measurements are done during this time.
  Value of the post-tetanus count at the time of administration of an extra bolus of rocuronium and the number of muscle contractions in response to a four-train stimulation
Characteristics of decurarization during spontaneous recovery phase | Usefulness of non depolarizing muscle relaxant-induced muscle paralysis is limited at the surgery period and should be avoided once the surgery is completed. Therefore, all measurements are done during this time.
  Delay of the gear ratio from train of four to 25; 75 and 90%.
When the TOF ratio will be greater than 0.9 on the TOF Watch side, the degree of residual paralysis will be assessed on the ITF side using 100 Hz tetanus stimulation repeated 5 times at 2 minutes interval | Usefulness of non depolarizing muscle relaxant-induced muscle paralysis is limited at the surgery period and should be avoided once the surgery is completed. Therefore, all measurements are done during this time.
  The response of theses tetanus stimulations will be compared with the one observed before myorelaxant administration but after induction of anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided